CLINICAL TRIAL: NCT03384420
Title: A Phase I/II, Open Label, Single Dose Clinical Study to Evaluate the Safety and Therapeutic Effects of Transplantation of MNV-BM-BLD (Autologous cd34+ Cells Enriched With Blood Derived Mitochondria) in Pediatric Patients With Pearson Syndrome
Brief Title: A Study to Evaluate the Safety and Therapeutic Effects of Transplantation of MNV-BM-BLD in Pediatric Patients With Pearson Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minovia Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNV-BM-BLD-001-IL
Record Dates: First submitted 2017-11-30; First posted 2017-12-27 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2020-06

CONDITIONS: Mitochondrial Diseases; Pearson Syndrome
Keywords: Autologous stem cell transplantation; Mitochondrial Diseases; Pearson Syndrome; Rare Diseases
MeSH Terms: conditions — Mitochondrial Diseases; VLCAD deficiency; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention CD34+ cells enriched with MNV-BLD (Experimental): Intervention CD34+ cells enriched with MNV-BLD
  Interventions: Biological: CD34+ cells enriched with MNV-BLD

INTERVENTIONS:
Biological: CD34+ cells enriched with MNV-BLD — Transplantation of autologous stem cell enriched with MNV-BLD (blood-derived mitochondria)

SUMMARY:
Mitochondrial diseases are a genetically heterogeneous group of disorders caused by mutations or deletions in mitochondrial DNA (mtDNA) displaying a wide range of severity and phenotypes. These diseases may be inherited from the mother (mitochondrial inheritance) or non-inherited. The latter are ultra-rare pediatric diseases caused by a mutation or deletion of mtDNA, which develop into a systemic multi organ disease and eventually death. MNV-BM-BLD is a therapeutic process for enrichment of patient's peripheral hematopoietic stem cells with normal and healthy mitochondria derived from donor blood cells. The process, called mitochondria augmentation therapy, aims to reduce the symptoms of mitochondrial diseases.

ELIGIBILITY:
Inclusion Criteria

1. Patient diagnosed with Pearson Syndrome, as verified by molecular identification of a defect in the mitochondrial DNA.
2. Normal maternal mitochondria as verified by mtDNA sequencing.
3. Males and females between 3 years or older and up to 18th birthday.
4. Patient is transfusion independent.
5. Patient has at least one of the following systematic involvements:

   1. High baseline lactate levels
   2. Episodes of metabolic crisis in the last year before pre-screening
   3. Renal failure (not dependent on dialysis) or evidence of proximal tubulopathy
   4. Growth retardation or failure to thrive

Exclusion Criteria

1. Absence of detectable mitochondria mutation or deletion.
2. Patient or patient's mother have a positive test for microbiologic
3. Patient is unable to undergo leukapheresis.
4. Patient suffers from chronic severe infection, malignant disease or any other disease or condition that may risk the patient or interfere with the ability to interpret the study results.
5. Patient has been treated previously with any cell or gene therapy.
6. Patient has participated in another clinical treatment trial or received other experimental medications outside of a clinical trial within 1 month prior to start of this study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-related adverse events as assessed by CTCAE v5.0 following MNV-BM-BLD during a follow up period of 12 months post treatment. | 1 year
  Severity will graded according to CTCAE, Version 5.0
IPMDS (International Pediatric Mitochondrial Disease Scale) | 1 year
  To compare the change in International Pediatric Mitochondrial Disease Scale (IPMDS) score during a follow up period of 12 months post treatment. IPMDS total score ranges from 0 to 243. The score is expressed as the percentage of items which were feasible to perform. The lower the score is, the higher the child's function

SECONDARY OUTCOMES:
Weight | 1 year
  To compare the changes (kilograms) to Baseline
Quantification of levels of normal mtDNA in blood and urine | 1 years
  To compare the changes to Baseline
Metabolic crisis events occurrence compared to two years prior to the study. | 3 Years
  To compare the changes during 3 years (2 years prior the study entry and 1 year follow up)
Change in renal function | 1 year
  Measurement of blood creatinine in a serum sample
Change in Brain involvement | 1 year
  Lactate peak as assessed by MRS
Height | 1 year
  To compare the changes (in meters) to Baseline
Change in cardiac function | 1 year
  Assessment of left ventricular ejection fraction via echocardiography
Monitoring for liver disease | 1 year
  Measurement of Aspartate Aminotransferase and Alanine aminotransferase level

OTHER OUTCOMES:
Hospitalization events | 1 year
  To compare the changes from medical history to 1 year follow up
Change in functional status | 1 year
  Distance traveled during the 6MWT (meters)
Change in hematological parameter | 1 year
  Measurement of hemoglobin level
Change in hematological parameter | 1 year
  Measurement of absolute neutrophil count
Change in hematological parameter | 1 year
  Measurement of platelet count
Control of blood glucose concentration | 1 year
  Hemoglobin A1c% in whole blood
ATP content. | 1 year
  To compare the changes to Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center Hospital- Tel Hashomer, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided